CLINICAL TRIAL: NCT02857881
Title: Effect of Simple Corneal De-epithelization Associated With a Therapeutic Photokeratectomy in Patients With Evolutive Keratoconus
Brief Title: Corneal De-epithelization Associated With a Therapeutic Photokeratectomy in Patients With Evolutive Keratoconus
Acronym: KERADES
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulty of inclusion of patients, impossible to reach the expected number
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ASD_2014-12
Record Dates: First submitted 2016-08-03; First posted 2016-08-05 (Estimated); Last update posted 2019-06-11 (Actual); Status verified 2019-06

CONDITIONS: Keratoconus
Keywords: keratoconus; photokeratectomy; de-epithelization
MeSH Terms: conditions — Keratoconus

ARMS (1):
- Evolutive keratoconus (Experimental)
  Interventions: Procedure: De-epithelization and therapeutic photokeratectomy

INTERVENTIONS:
Procedure: De-epithelization and therapeutic photokeratectomy

SUMMARY:
Keratoconus is a symmetrical, bilateral, non-inflammatory, idiopathic corneal pathology, characterized by a progressive corneal thinning. This disease leads to a bombing of the cornea, inducing a strong corneal astigmatism, responsible for a loss of visual acuity sometimes very important, non-correctable by lens of glasses. Collagen Cross-Linking (CXL) and simple corneal de-epithelization are two common surgical technics aiming to slow the progression of this pathology. They consist in rigidifying the corneal structure in order to stabilize its deformation progression. Even though these technics are commonly performed, none of these strategies has proven their efficiency. The effects of CXL can be due to the superficial scarring reaction as well as the effects of corneal remodeling induced by the de-epithelization phase during a CXL procedure, and not due to the covalent links between collagen and fibrils, formed by the biochemical reaction resulting from the UV-A exposition in the presence of Riboflavine De-epithelization may be an equally effective treatment, when compared to CXL, but without long term secondary effects. Its association with a therapeutic photokeratectomy (PKT, surgical technic used to regulate the corneal surface, and eliminate its opacities in order to recuperate the transparency of the cornea) will aim to improve the regularity of the anterior corneal surface, thus allowing a better epithelial attachment (adhesion) and may allow a stromal inflammatory reaction, favorable to the improvement of corneal biomechanics. PKT is a reliable technic; however it has not yet proven its efficiency in the treatment of keratoconus.

The purpose of this study is to describe the effects of de-epithelization associated with a therapeutic photokeratectomy in patients with evolutive keratoconus, by showing the proportion of patients who lost the evolutivity of their keratoconus, after 6 months and 1 year, after an intervention of de-epithelization associated with therapeutic photokeratectomy.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged from 15 to 45 years old
* Patients with an evolutive keratoconus
* Planned intervention (de-epithelization and photokeratectomy)

Exclusion Criteria:

* Contra-indication to de-epithelization (active scarring corneal lesion)
* Pregnant women and breastfeeding
* Absence of the written consent to participate in the trial

Ages: 15 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2015-10-13 (Actual); Primary Completion 2019-02-07 (Actual); Study Completion 2019-02-07 (Actual)

PRIMARY OUTCOMES:
Evolutivity of keratoconus (Proportion of patients who lost the evolutivity of their keratoconus) | 6 months
  Effects of de-epithelization associated with a therapeutic photokeratectomy in patients with evolutive keratoconus, by showing the proportion of patients who lost the evolutivity of their keratoconus, after 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Fondation Ophtalmologique Adolphe de Rothschild, Paris, France